CLINICAL TRIAL: NCT04265183
Title: Preformed Metal Crowns (PMCs) as a Treatment of Children With Hypomineralised Second Primary Molars (HSPM) Using the Hall Technique (HT)
Brief Title: PMCs as a Treatment of Children With HSPM Using the HT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Emily Mampay, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B322201837979
Record Dates: First submitted 2020-01-20; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hypomineralization of Enamel
Keywords: preformed metal crowns; Hall technique
MeSH Terms: conditions — Dental Enamel Hypomineralization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients treated with preformed metal crowns (Experimental): All patients included received a preformed metal crown on their HSPM affected teeth.
  Interventions: Other: Placing preformed metal crowns using Hall technique.

INTERVENTIONS:
Other: Placing preformed metal crowns using Hall technique. — Preformed metal crowns (3M™ ESPE™ STAINLESS STEEL CROWNS) were placed after using separation elastics (Dentalastics® separators, DENTAURUM). The crowns were cemented using is a self-curing, radiopaque, fluoride-releasing, resin-modified glass ionomer luting cement (Ketac™ Cem Plus Luting Cement, 3M™ ESPE™). The technique used to place the crowns was the Hall technique (technique without tooth preparation).

SUMMARY:
Hypomineralised primary second molars are primary molars with a developmental disorder of the enamel. Preformed metal crowns already have good results for the treatment of caries on primary molars. In this study the aim is to investigate the clinical success and overall survival of preformed metal crowns as a treatment for hypomineralised primary molars. The crowns were placed using the Hall technique which is a simplified way of placing these crowns.

ELIGIBILITY:
Inclusion Criteria:

* age 2-12 years
* American Society of Anesthesiologists(ASA)-score I: healthy patient
* hypomineralisation grade: 2-6
* caries with an International Caries Detection and Assessment System (ICDAS)- score: 0-3
* limited provoked pain complaint

Exclusion Criteria:

* caries with an ICDAS-score: 4-6
* pulpitis pain complaints
* infection (clinical and/or radiographic)
* >1/3 root resorption
* allergies to the used materials

Ages: 24 Months to 144 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
The clinical success of preformed metal crowns using Hall technique on hypomineralised second primary molars based on clinical acceptable results. | 1-2 year
  The results are clinical acceptable when there are no clinical signs of infection of the tooth, no caries development or heavy bleeding of the gingiva (after probing).
The overall survival rate of preformed metal crowns using Hall technique on hypomineralised second primary molars is defined as acceptable clinical outcomes. | 1-2 year
  The outcomes are clinically acceptable when there are no signs of infection (abscess) or caries.
The overall survival rate of preformed metal crowns using Hall technique on hypomineralised second primary molars is defined as acceptable radiographical outcomes. | 1-2 year
  The outcomes are radiographical acceptable when no signs of infection or interproximal bone loss are seen on the radiographs.

SECONDARY OUTCOMES:
The results can be affected by bruxism. Signs of bruxism will not mean failure. We will rate the wear as acceptable or successful. This bruxism will be measured by clinical signs of wear on the crowns. | 1-2 year
  When the wear of the crown is limited to minimal loss of metal, it is rated successful. When the wear is going through the full thickness of the crown until the underlying tooth structure, it is rated as acceptable.
The oral hygiene of the patient will be measured using the Simplified Oral Hygiene Index. The minimum value is 0: clean. The maximum value is 3: tooth surface covered with >2/3 soft dental plaque. The higher the score, the worse the outcome. | 1-2 year
  Oral hygiene of the patients scored as debris >1/3 of the crown surface is scored as bad oral hygiene. Bad oral hygiene implies a higher prevalence of (heavy) bleeding of the gingiva after probing. Which has a significant influence on the clinical success of the crowns.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Declerck, Prof. Dr., Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayhew D, Mendonca V, Murthy BVS. A review of ASA physical status - historical perspectives and modern developments. Anaesthesia. 2019 Mar;74(3):373-379. doi: 10.1111/anae.14569. Epub 2019 Jan 15. PMID 30648259
- [Background] Ghanim A, Elfrink M, Weerheijm K, Marino R, Manton D. A practical method for use in epidemiological studies on enamel hypomineralisation. Eur Arch Paediatr Dent. 2015 Jun;16(3):235-46. doi: 10.1007/s40368-015-0178-8. Epub 2015 Apr 28. PMID 25916282
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Kulkarni P, Agrawal S, Bansal A, Jain A, Tiwari U, Anand A. Assessment of nickel release from various dental appliances used routinely in pediatric dentistry. Indian J Dent. 2016 Apr-Jun;7(2):81-5. doi: 10.4103/0975-962X.184649. PMID 27433051
- [Result] Tonmukayakul U, Martin R, Clark R, Brownbill J, Manton D, Hall M, Armfield J, Smith M, Shankumar R, Sivasithamparam K, Martin-Kerry J, Calache H. Protocol for the Hall Technique study: A trial to measure clinical effectiveness and cost-effectiveness of stainless steel crowns for dental caries restoration in primary molars in young children. Contemp Clin Trials. 2015 Sep;44:36-41. doi: 10.1016/j.cct.2015.07.005. Epub 2015 Jul 18. PMID 26196586
- [Result] Wada K, Kanazawa H, Kudo M, Kindaichi J, Miyashin M. Management of developmental enamel defects in the primary dentition. J Oral Sci. 2017;59(3):457-460. doi: 10.2334/josnusd.16-0805. PMID 28904324
- See also: Restorative management of dental enamel defects in the primary dentition — https://doi.org/10.1007/s41894-018-0040-6